CLINICAL TRIAL: NCT06059417
Title: Foam Tape Allergy a Sticky Situation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHRISTUS Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-009
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Medical Adhesive Allergy; Dermatologic Conditions; Dermatologic Lesions
Keywords: Dermatology; Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: A cohort of consenting, healthy physicians, nurses, and ancillary staff at a teaching facility who did not have known hypersensitivity to foam tape were enrolled. Study investigators applied a 2x2 inch piece of 3M micro-foam adhesive to the medial aspect of each subject's upper arm. The contralateral arm served as a reference for comparison. The adhesive remained in place for 48 hours and the study authors assessed patients utilizing the previously validated Cutaneous Irritancy Scoring System (CISS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foam-tape/Control (Other): One of the participants upper extremity (arm) was used for intervention and the same participants other arm was used as the control in this study.
  There was only 1 research arm in this study and all study participants were in it.
  Interventions: Other: 2x2 inch piece of 3M microfoam adhesive

INTERVENTIONS:
Other: 2x2 inch piece of 3M microfoam adhesive — A 2x2 inch piece of 3M microfoam adhesive will be applied to the medial aspect of the subject's upper arm.
  The adhesive will remain in place for 48 hours at which time an investigator will remove the adhesive and assess the study area. A numerical value will be assigned based on the Cutaneous Irritancy Scoring System (CISS). The study site will be compared to the contra-lateral upper extremity at the end of the 48 hour period.

SUMMARY:
Foam tape is commonly used in the emergency department as a dressing over chest tubes owing to its occlusive and compressible properties. There is a paucity of data regarding the incidence of significant cutaneous reactions to this material. The investigators conducted a prospective trial to evaluate the incidence of dermatitis following application of foam tape to the upper arm of a cohort of healthy volunteers.

DETAILED DESCRIPTION:
This was a prospective, interventional trial. The investigators enrolled a cohort of consenting, healthy physicians, nurses, and ancillary staff at a teaching facility who did not have known hypersensitivity to foam tape. Study investigators applied a 2x2 inch piece of 3M micro-foam adhesive to the medial aspect of each subject's upper arm. The contralateral arm served as a reference for comparison. The adhesive remained in place for 48 hours and the study authors assessed patients utilizing the previously validated Cutaneous Irritancy Scoring System (CISS). Categorical variables analyzed by chi-square, continuous variables with t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70
* No reported history of dermatologic conditions
* No active dermatologic lesions
* Able to provide written consent to participation in the study.
* Resident and/or ancillary staff

Exclusion Criteria:

* Hospitalized patients
* Adults unable to consent.
* Prisoners
* Adults with anaphylaxis to medical adhesives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Cutaneous Irritancy Scoring System | 48 hours
  A score will be assigned to the test area using the established Cutaneous Irritancy Scoring System. Using an established scoring system grading based on erythema and edema, a cumulative score will be obtained by adding erythema and edema. A score of 0 is no reaction. A score of 1-3 is mild, 4-5 is moderate, and 6-8 severe.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CHRISTUS Health/Texas A&M Health Science Center, Corpus Christi, Texas
  - CHRISTUS Health, Corpus Christi, Texas

REFERENCES:
- [Result] Smith SM, Zirwas MJ. Nonallergic reactions to medical tapes. Dermatitis. 2015 Jan-Feb;26(1):38-43. doi: 10.1097/DER.0000000000000098. PMID 25581669
- [Result] Widman TJ, Oostman H, Storrs FJ. Allergic contact dermatitis from medical adhesive bandages in patients who report having a reaction to medical bandages. Dermatitis. 2008 Jan-Feb;19(1):32-7. PMID 18346394
- [Result] Dykes PJ. The effect of adhesive dressing edges on cutaneous irritancy and skin barrier function. J Wound Care. 2007 Mar;16(3):97-100. doi: 10.12968/jowc.2007.16.3.27013. PMID 17385583
- [Result] Wood MD, Powers J, Rechter JL. Comparative Evaluation of Chest Tube Insertion Site Dressings: A Randomized Controlled Trial. Am J Crit Care. 2019 Nov;28(6):415-423. doi: 10.4037/ajcc2019645. PMID 31676515
- [Derived] Vo NH, Richman P, Torres R, Xu KT, Miller M. The incidence of dermatitis following application of foam tape in healthy volunteers-A prospective trial. Am J Emerg Med. 2024 May;79:212-213. doi: 10.1016/j.ajem.2024.02.043. Epub 2024 Mar 5. PMID 38462426